CLINICAL TRIAL: NCT01679938
Title: Prevention of Obesity in Children: An Intervention Based on Child Care Centers Belonging to the Mexican Institute of Social Security
Brief Title: A Child Care-based Obesity Prevention Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Salud Publica, Mexico (Other)
Collaborators: National Council of Science and Technology, Mexico (Other); Instituto Mexicano del Seguro Social (Other Government); Harvard Pilgrim Health Care (Other)
Responsible Party: Principal Investigator, Hortensia Reyes Morales, Principal Investigator, Instituto Nacional de Salud Publica, Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SALUD-2009-01-114027
Record Dates: First submitted 2012-08-24; First posted 2012-09-06 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Obesity
Keywords: obesity prevention; cluster-randomized controlled trial; preschool-aged children
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- primary obesity prevention (Experimental): The intervention will involve four main components:
  1. Training of child care providers.
  2. Curriculum sessions for children.
  3. Family outreach activities.
  4. Maintenance activities.
  Interventions: Behavioral: primary obesity prevention
- Control group (No Intervention): For the control group, usual care will be provided

INTERVENTIONS:
Behavioral: primary obesity prevention — 1. Training of child care providers.
  2. Curriculum sessions for children. Child care providers will facilitate 12 interactive education sessions that focus on key obesity-related behaviors.
  3. Family outreach activities. Child care providers and research staff will communicate behavior change messages to families through ten take-home activities focused on key obesity-related behaviors and through monthly family workshops at the child care center.
  4. Maintenance activities. Over the six months following the main intervention, research staff will conduct eight booster sessions for the children and one booster session for the family that will build upon activities and behavior change messages of the main intervention.
  Arms: primary obesity prevention

SUMMARY:
The overall objective is to determine the impact of comprehensive, multifaceted, child care-based intervention to prevent obesity among children 2 through 5 years of age. The specific aims are:

1. To determine the extent to which the intervention, compared with the control condition, results in a smaller age-associated increase in body mass index (BMI) after a 6-month intervention (primary outcome) and a 1-year follow-up period among children.
2. To determine the extent to which the intervention, compared with the control condition, reduces the proportion of children who are obese (BMI >95th percentile for age and sex).
3. To determine the extent to which the intervention, compared with the control condition, results in:

   1. improved dietary, physical activity and television-viewing behaviors among children, specifically, reducing the consumption of sugar-sweetened beverages, high calorie/low nutrient-dense snack foods, and fast food, increasing active time, and reducing TV/video viewing time;
   2. improved home food and activity environment, specifically, decreasing availability of sugar-sweetened beverages and high calorie/low nutrient-dense snack foods, and increasing parental support for healthy eating and regular physical activity;
   3. improved child care center food and activity environment, specifically, increasing opportunities for healthy eating and physical activity, and increasing support and encouragement of children's behavior change by child care providers;
4. To assess the feasibility and acceptability of the intervention among child care providers and families.

METHODS. The investigators will conduct a cluster-randomized controlled trial in 16 IMSS child care centers in Mexico City. The investigators will randomly assign 8 child care centers to the intervention condition and 8 to an assessment-only control condition.

Multifaceted intervention. The resulting intervention will involve four main components:

1. Training of child care providers.
2. Curriculum sessions for children.
3. Family outreach activities.
4. Maintenance activities. Outcome and process measurements. Age-associated BMI (child's), changes in child's key obesity-related behaviors, changes in the child's home food and activity environment, and changes in child care food and activity environment. At the intervention and control child care sites, changes from baseline to one year for all outcome variables will be measured.

DETAILED DESCRIPTION:
Over the past 20 years, the prevalence of obesity in Mexico has increased dramatically among individuals across the lifespan, including even the youngest populations.National data from the Mexican Institute of Social Security (IMSS) population estimate that nearly 15% of children aged 2 to 5 years are obese as defined by World Health Organization criteria. Obesity among preschool-aged children is of serious public health concern due to its adverse effects on children's physical and psychosocial well-being,and its association with obesity risk in later childhood, adolescence, and young adulthood. Furthermore, because dietary and activity patterns have not been firmly established, early childhood represents a critical window for prevention.

Given the high number of preschool children enrolled in out-of-home child care in Mexico, important opportunities exist for developing child care-based obesity prevention interventions focused on promoting healthy activity and dietary behaviors among children. Child care centers provide an ideal setting for a multi-level, ecologic intervention that includes strategies aimed at environmental level changes within the child care center, as well as individual level behavior change among the children. In addition, child care-based interventions have the potential to reach out to the children's families to improve the child's home food and activity environment.

Setting and study population. There are 142 IMSS child care centers in Mexico City. To allow for adequate attention to details in the development of the intervention and evaluation protocol and to contain costs prior to broad dissemination of the program, the investigators will focus on 16 IMSS child care sites for this proposal, which together provide care for approximately 450 children aged 2 to 5 years. At each IMSS child care center a team consisting of a nutritionist, a nurse, an educator, and child care technicians provides the daily care and education programs for the children. This extensive personnel structure provides the ideal infrastructure for implementing the proposed multifaceted intervention.

Since the intervention is a primary prevention program, the investigators will make the program available to all children, aged 2 to 5 years, at the child care centers, regardless of their current weight status. Children with chronic conditions that limit ability to measure height and weight or substantially interfere with growth, physical activity, or dietary recommendations will be excluded.

Data analysis for outcome measures. Intent-to-treat analyses to compare study outcomes between the intervention and control groups at post-intervention and at 6-months follow-up will be used. To compare the difference the age-associated increase in body mass index (BMI) among intervention and control groups (Aim 1), the mixed effects model with group (child care center) as the clustering factor will be used, as recommended by several authoritative sources. Similar analyses to compare the difference in prevalence of overweight (Aim 2), in the children's weight-related behaviors (Aim 3a), in the children's home environment (Aim 3b), and in the environment of the child care center (Aim 3c) will be performed.

ELIGIBILITY:
Inclusion Criteria:

* IMSS child care centers with at least 40 children aged 2-4 years
* Child care center director that is willing to participate in the study and agrees to be randomized to control or intervention conditions. Since the intervention is a primary prevention program, the program will be available to all children, aged 2 to 4 years, at the child care centers, regardless of their current weight status
* Children's parents who sign a consent form indicating their permission for their child to participate in the study and their willingness to participate in the measurement activities

Exclusion Criteria:

* Children with chronic conditions that limit ability to measure height and weight or substantially interfere with growth, physical activity, or dietary recommendations from the measurement activities

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 640 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2012-11 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Child's age-associated Body Mass Index | Change from baseline (May 2011) at one year follow-up (November 2012)
  The investigators will measure standing height for all participants over the age of 3 years, and from 2-3 years when possible. For some participants between age 2 and 3 years requiring recumbent lengths, a recumbent board and the recumbent to standing correction factor recommended by the U.S. Centers for Disease Control and Prevention (0.8 cm)will be used.In all cases, BMI will be the ratio of weight (kg) to the square of standing height (m). Accepted definition of obese (BMI >95th percentile for age and sex) and overweight (BMI 85th - 95th percentile for age and sex)will be used. All height and weight measurements will be conducted in a private area at the child care sites.

SECONDARY OUTCOMES:
Children's home environment | Change from baseline at one year follow-up.
  To assess the home food and nutrition environment, research staff will conduct in-person surveys with parents using items from the Healthy Home Survey. The Healthy Home Survey was designed to assess key aspects of the diet and activity home environment, including availability of foods, role modeling by parents of behaviors, and parental support for healthy behaviors.
Children's key obesity-related behaviors. | Change from baseline at one year of follow-up.
  Research staff will conduct brief, in-person surveys with parents to measure children's obesity-related behaviors. The in-person surveys will include questions about the children's behaviors and the children's home dietary and activity environment and will be conducted at the child care center when parents come to pick up their children.

CONTACTS AND LOCATIONS:
Overall Officials: Hortensia Reyes-Morales, DrSc, Principal Investigator — Instituto Nacional de Salud Publica, Mexico
Locations (1):
- Instituto Nacional de Salud Pública, Cuernavaca, Morelos, Mexico

REFERENCES:
- [Result] Rodriguez-Oliveros G, Haines J, Ortega-Altamirano D, Power E, Taveras EM, Gonzalez-Unzaga MA, Reyes-Morales H. Obesity determinants in Mexican preschool children: parental perceptions and practices related to feeding and physical activity. Arch Med Res. 2011 Aug;42(6):532-9. doi: 10.1016/j.arcmed.2011.10.006. Epub 2011 Oct 21. PMID 22019411